CLINICAL TRIAL: NCT04872803
Title: Emotional Security and Quality of Life Among Breast Cancer Patient Who Have Undergo Mastectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Omar, Assistant Lecturer, Assiut University
Other Study IDs: Emotional security&mastectomy
Record Dates: First submitted 2021-04-27; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Mastectomy
Keywords: Mastectomy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common cause of cancer death among women worldwide. Incidence rates are high in more developed countries than rates in less developed countries In Egypt, standardized age of cancers are 166.6per 100.000 in both sexes cancer breast represent 32%in females and 15.4%in both sexes of all cancer Mastectomy is an important treatment method in Brest cancer. But, mastectomy has a deep and stable negative impact on a woman because, mastectomy as a treatment option, can result in a sense of mutilation and diminished self-worth and may threaten perceptions of femininity Body image of a woman includes the symbolic meaning and importance of her breasts. The more she values her breasts, more devastating effects of having a mastectomy can be. it has been reported that cutting off/amputating one or both breasts was associated with several problems in women such as loss of fertility, charm and sexuality, fear of recurrence Social support plays an important role in reducing the pressure and improving health. Cancer patients who lack social support may be more pessimistic and desperate as they are constantly looking for support from others Therefore, it is critical for health care professionals to become familiar with the impact of a breast cancer diagnosis and its treatment on patient's quality of life .

DETAILED DESCRIPTION:
Breast cancer is the most common cause of cancer death among women worldwide. Incidence rates are high in more developed countries than rates in less developed countries In Egypt, standardized age of cancers are 166.6per 100.000 in both sexes cancer breast represent 32%in females and 15.4%in both sexes of all cancer Mastectomy is an important treatment method in Brest cancer. But, mastectomy has a deep and stable negative impact on a woman because, mastectomy as a treatment option, can result in a sense of mutilation and diminished self-worth and may threaten perceptions of femininity Body image of a woman includes the symbolic meaning and importance of her breasts. The more she values her breasts, more devastating effects of having a mastectomy can be. it has been reported that cutting off/amputating one or both breasts was associated with several problems in women such as loss of fertility, charm and sexuality, fear of recurrence Social support plays an important role in reducing the pressure and improving health. Cancer patients who lack social support may be more pessimistic and desperate as they are constantly looking for support from others Therefore, it is critical for health care professionals to become familiar with the impact of a breast cancer diagnosis and its treatment on patient's quality of life

ELIGIBILITY:
Inclusion Criteria:

1. female patient between 18y and 55y
2. a first-time breast cancer diagnosis
3. post-operative mastectomized patients
4. clear consent to participate in study

Exclusion Criteria:

1. male gender
2. females patient with concurrent comorbid psychiatric or neurological disorders
3. age younger than 18y
4. patients with disease recurrence, patients presenting with other malignancies

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female patient between 18y and 55y with first-time breast cancer diagnosis and post-operative mastectomized patients
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life post mastectomy | 6 months
  To evaluate the impact of breast cancer on the quality of life

SECONDARY OUTCOMES:
Stages of breast cancer and emotional security | 6 months
  Studying the effect of different stages of breast cancer and its duration on the emotional security

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Omar, Master, Principal Investigator — Assiut University